CLINICAL TRIAL: NCT01003015
Title: An Uncontrolled Open Label Multicenter Phase II Safety Study of BAY73-4506 in Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Safety Study of BAY73-4506 in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14596; 2009-012570-13 (EudraCT Number)
Record Dates: First submitted 2009-10-02; First posted 2009-10-28 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; Safety; BAY73-4506
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY73-4506

INTERVENTIONS:
Drug: BAY73-4506 — 160 mg BAY73-4506

SUMMARY:
The purpose of this study is to determine whether BAY73-4506 treatment is safe and can shrink or delay the growth of tumors in patients with unresectable liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged equal or above 18 years.
* BCLC stage Category A, B or C that cannot benefit from treatments of established efficacy with higher priority such as resection, liver transplantation, local ablation, chemoembolization or systemic sorafenib.
* Liver function status Child-Pugh class A.
* Failure to prior treatment with sorafenib (defined as radiological progression under sorafenib therapy)
* Local or loco-regional therapy (eg, surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed = 4 weeks before first dose of BAY73-4506.
* ECOG PS of 0 or 1.
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Prior systemic treatment with molecular targeted agents for HCC, except sorafenib. Prior chemotherapy treatment is allowed.
* Known history or symptomatic metastatic brain or meningeal tumors (head CT or MRI at screening to confirm the absence of central nervous system [CNS] disease if patient has symptoms suggestive or consistent with CNS disease).
* Congestive heart failure NYHA>/= class 2
* Unstable angina (angina symptoms at rest, new onset angina within the last 3 months) or myocardial infarction (MI) within the past 6 months before start of study medication.
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Adverse Event Collection | Up to 30+/- 7 days after permanently discontinuing BAY73-4506 administration

SECONDARY OUTCOMES:
Time to progression | Every 6 weeks during treatment and after 6 cycle treatment every 18 weeks till progression
Objective response rate | Every 6 weeks during treatmen and after 6 cycle treatment every 18 weeks till progression
Disease control rate | Every 6 weeks during treatmen and after 6 cycle treatment every 18 weeks till progression
Overall survival | Every 6 weeks during treatmen and after 6 cycle treatment every 18 weeks till progression
Trough concentration of Regorafenib and metabolites (for Europe only) | Cycle 1 Day 15 and Cycle 2 Day 1
Full Pharmacokinetics profile of BAY73-4506 and metabolites (for Korea only) | Cycle 1 Day 21 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- Germany (5):
  - Regensburg, Bavaria
  - Frankfurt am Main, Hesse
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Magdeburg, Saxony-Anhalt
- Italy (4):
  - Rozzano, Milano
  - Bologna
  - Milan
  - Roma
- South Korea (2):
  - Daegu
  - Seoul
- Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Bruix J, Tak WY, Gasbarrini A, Santoro A, Colombo M, Lim HY, Mazzaferro V, Wiest R, Reig M, Wagner A, Bolondi L. Regorafenib as second-line therapy for intermediate or advanced hepatocellular carcinoma: multicentre, open-label, phase II safety study. Eur J Cancer. 2013 Nov;49(16):3412-9. doi: 10.1016/j.ejca.2013.05.028. Epub 2013 Jun 25. PMID 23809766